CLINICAL TRIAL: NCT00032591
Title: CSP #481 - The Home INR Study (THINRS)
Brief Title: The Home INR Study
Acronym: THINRS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 481
Record Dates: First submitted 2002-03-27; First posted 2002-03-28 (Estimated); Results first posted 2014-02-06 (Estimated); Last update posted 2014-04-15 (Estimated); Status verified 2014-03

CONDITIONS: Atrial Fibrillation
Keywords: AF; Mechanical heart valve (MHV)
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Active Comparator): Patient Self-Testing (PST) of prothrombin time by international normalized ratio (PT-INR or INR) with weekly testing
  Interventions: Procedure: Weekly patient self-testing of prothrombin time
- Arm 2 (Other): High quality anticoagulation management (HQACM) with conventional monthly testing
  Interventions: Other: High quality anticoagulation management (HQACM) with conventional monthly testing

INTERVENTIONS:
Procedure: Weekly patient self-testing of prothrombin time
  Arms: Arm 1
Other: High quality anticoagulation management (HQACM) with conventional monthly testing — HQACM with testing every 4 weeks and as indicated for out of range values, medication/clinical changes.
  Other Names: HQACM
  Arms: Arm 2

SUMMARY:
Since home monitors of prothrombin time (PT) may potentially improve the safety, quality, and convenience of chronic anticoagulation management, it is likely that there will be demands from providers, patients, and manufacturers to make home monitors available to VA patients. The rationale for patient self-testing (PST) is that, compared to conventional high quality anticoagulation management (HQACM), it would permit more intense monitoring and increased patient participation in his/her own care, resulting in increased precision in anticoagulation control and thus fewer events of thromboembolism (strokes) and bleeding. The secondary hypothesis is that PST and HQACM will be comparable in terms of health care utilization and cost.

DETAILED DESCRIPTION:
Intervention: Weekly patient self-testing (PST) of prothrombin time by international normalized ratio (PT INR) versus conventional monthly high quality anticoagulation management (HQACM) from an anticoagulation clinic with a minimum two years follow-up.

Primary Hypothesis: Compared to conventional monitoring in the clinic, PST of anticoagulation intensity will decrease the number of events of thromboembolism (strokes), bleeding, and all cause deaths and improve the quality of anticoagulation.

Second Hypothesis: PST and conventional monitoring will be comparable in terms of health care utilization and cost.

Primary Outcomes: Event rates (thromboembolism or bleeding episodes), time to first event, time within therapeutic range for anticoagulation intensity, and total health care cost (including price of PST monitors) and utilization.

Study Abstract: Since home monitors of prothrombin time (PT) may potentially improve the safety, quality, and convenience of chronic anticoagulation management, it is likely that there will be demands from providers, patients, and manufacturers to make home monitors available to VA patients. The rationale for PST is that it would permit more intense monitoring and increased patient participation in his/her own care, resulting in increased precision in anticoagulation control and thus fewer events.

Original plan was for a study at 32 sites with a total sample size of about 3,200 patients and a length of three years (one for recruitment and two years of follow-up). Final status was 28 sites that randomized 2922 patients in 2.75 years of recruitment with a minimum of two years of follow-up.

ELIGIBILITY:
Inclusion Criteria:

To be enrolled in this study, patients must:

1. have AF and/or a MHV;
2. be scheduled to receive warfarin indefinitely (operationally defined as 2 years);
3. be using warfarin according to the criteria described in the Coumadin package insert (no off-label uses);
4. be expected to survive for the duration of the study;
5. not be suffering from intracranial bleeding (intracranial hemorrhage, subarachnoid hemorrhage, hemorrhagic stroke) or any other contraindication described in the Coumadin package insert;
6. be willing to perform PST;
7. be willing to be randomized;
8. possess adequate cognitive and language skills to follow the protocol and all related instructions;
9. be willing to participate for the full duration of the study;
10. sign the informed consent form; and
11. not be enrolled in another randomized clinical trial that involves a drug or device intervention.

Exclusion Criteria:

Patients are excluded in this study if:

1. subject has had intracranial hemorrhage, subarachnoid hemorrhage, hemorrhagic stroke, or any other absolute/major contraindication described in the warfarin package insert within the last month
2. subject enrolled in another randomized clinical trial that involves a drug or device intervention
3. subject is not able to follow the protocol and all related instructions, and does not have a caregiver with these skills

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2922 (Actual)
Dates: Start 2003-08; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David B. Matchar, MD, Study Chair — Durham VA Medical Center HSR&D COE
Locations (29):
- United States (28):
  - VA Medical Center, Birmingham, Birmingham, Alabama
  - VA Central California Health Care System, Fresno, Fresno, California
  - VA Medical Center, Loma Linda, Loma Linda, California
  - VA Palo Alto Health Care System, Palo Alto, California
  - VA Greater Los Angeles Healthcare System, West LA, West Los Angeles, California
  - VA Eastern Colorado Health Care System, Denver, Denver, Colorado
  - VA Connecticut Health Care System (West Haven), West Haven, Connecticut
  - Edward Hines, Jr. VA Hospital, Hines, Illinois
  - VA Medical Center, North Chicago, North Chicago, Illinois
  - VA Medical Center, Iowa City, Iowa City, Iowa
  - VA Maryland Health Care System, Baltimore, Baltimore, Maryland
  - John D. Dingell VA Medical Center, Detroit, Detroit, Michigan
  - VA Medical Center, Minneapolis, Minneapolis, Minnesota
  - VA Medical Center, Kansas City MO, Kansas City, Missouri
  - Las Vegas, North Las Vegas, Nevada
  - VA Sierra Nevada Health Care System, Reno, Nevada
  - VA Western New York Healthcare System at Buffalo, Buffalo, New York
  - VA Medical Center, Syracuse, Syracuse, New York
  - VA Medical Center, Bronx, The Bronx, New York
  - Durham VA Medical Center HSR&D COE, Durham, North Carolina
  - VA Medical Center, Cleveland, Cleveland, Ohio
  - VA Medical Center, Oklahoma City, Oklahoma City, Oklahoma
  - VA Pittsburgh Health Care System, Pittsburgh, Pennsylvania
  - VA Medical Center, Providence, Providence, Rhode Island
  - VA North Texas Health Care System, Dallas, Dallas, Texas
  - VA South Texas Health Care System, San Antonio, San Antonio, Texas
  - VA Medical Center, Salem VA, Salem, Virginia
  - Wlliam S. Middleton Memorial Veterans Hospital, Madison, Madison, Wisconsin
- VA Medical Center, San Juan, San Juan, Puerto Rico

REFERENCES:
- [Result] Dolor RJ, Ruybalid RL, Uyeda L, Edson RG, Phibbs C, Vertrees JE, Shih MC, Jacobson AK, Matchar DB; THINRS Site Investigators. An evaluation of patient self-testing competency of prothrombin time for managing anticoagulation: pre-randomization results of VA Cooperative Study #481--The Home INR Study (THINRS). J Thromb Thrombolysis. 2010 Oct;30(3):263-75. doi: 10.1007/s11239-010-0499-8. PMID 20628787
- [Result] Matchar DB, Jacobson A, Dolor R, Edson R, Uyeda L, Phibbs CS, Vertrees JE, Shih MC, Holodniy M, Lavori P; THINRS Executive Committee and Site Investigators. Effect of home testing of international normalized ratio on clinical events. N Engl J Med. 2010 Oct 21;363(17):1608-20. doi: 10.1056/NEJMoa1002617. PMID 20961244
- [Result] Matchar DB, Jacobson AK, Edson RG, Lavori PW, Ansell JE, Ezekowitz MD, Rickles F, Fiore L, Boardman K, Phibbs C, Fihn SD, Vertrees JE, Dolor R. The impact of patient self-testing of prothrombin time for managing anticoagulation: rationale and design of VA Cooperative Study #481--the Home INR Study (THINRS). J Thromb Thrombolysis. 2005 Jun;19(3):163-72. doi: 10.1007/s11239-005-1452-0. PMID 16082603
- [Derived] Phibbs CS, Love SR, Jacobson AK, Edson R, Su P, Uyeda L, Matchar DB; writing for the THINRS Executive Committee and Site Investigators. At-Home Versus In-Clinic INR Monitoring: A Cost-Utility Analysis from The Home INR Study (THINRS). J Gen Intern Med. 2016 Sep;31(9):1061-7. doi: 10.1007/s11606-016-3700-8. Epub 2016 May 27. PMID 27234663
- [Derived] Matchar DB, Love SR, Jacobson AK, Edson R, Uyeda L, Phibbs CS, Dolor RJ. The impact of frequency of patient self-testing of prothrombin time on time in target range within VA Cooperative Study #481: The Home INR Study (THINRS), a randomized, controlled trial. J Thromb Thrombolysis. 2015 Jul;40(1):17-25. doi: 10.1007/s11239-014-1128-8. PMID 25209313

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment started in August 2003 and ended at the end of May 2006. Participating sites were VA Medical Centers with anticoagulation services with active rosters of more than 400 patients.
Pre-assignment Details: A total of 3745 participants were consented and screened. Out of this total, 823 were excluded from the study. The majority of those excluded is due to participants not doing or passing the competency assessment.
Groups:
- Patient Self-Testing (PST): Patient Self-Testing (PST) of prothrombin time by international normalized ratio (PT-INR or INR) with weekly testing
- High Quality Anticoagulation Management (HQACM): High quality anticoagulation management (HQACM) with conventional monthly testing
Period: Screening
Arm/Group | Patient Self-Testing (PST) | High Quality Anticoagulation Management (HQACM)
Started | 1873 (3745 patients provided informed consent and were screened for participation.) | 1872 (Treatment assigned at randomization; screening counts by arm represent half of the total screened.)
Completed | 1465 (823 were excluded from the study) | 1457
Not Completed | 408 | 415
Period: Randomization
Arm/Group | Patient Self-Testing (PST) | High Quality Anticoagulation Management (HQACM)
Started | 1465 (2922 underwent randomization) | 1457
Completed | 1465 (1465 were assigned to self-testing) | 1457 (1457 were assigned to clinic testing)
Not Completed | 0 | 0
Period: Follow-up
Arm/Group | Patient Self-Testing (PST) | High Quality Anticoagulation Management (HQACM)
Started | 1465 (2 were lost to follow-up, both with Atrial Fibrillation, no Mechanical Heart Valves) | 1457 (5 were lost to follow-up, all with Atrial Fibrillation, no Mechanical Heart Valves)
Completed | 1463 (1463 were included in analysis with greater than 1 day of follow-up) | 1452 (1452 were included in analysis with greater than 1 day of follow-up)
Not Completed | 2 | 5

BASELINE CHARACTERISTICS:
Population: 3745 participants were screened for participation
Groups:
- Total: Total of all reporting groups
Arm/Group | Patient Self-Testing (PST) | High Quality Anticoagulation Management (HQACM) | Total
Number analyzed (Participants) | 1465 | 1457 | 2922
Age, Continuous [Mean (Standard Deviation); unit: years]
  Total study population | 66.6 (9.7) | 67.4 (9.4) | 67 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 26 | 51
  Male | 1440 | 1431 | 2871

OUTCOME MEASURES:

1. Primary Outcome: Time to First Event (Death, Stroke, Major Bleed)
Description: Time to first event (death, stroke, major bleed)
  The primary outcome was time to first event, and we used the Kaplan-Meier method to compare survival curves and the results using the log-rank test. The number of patients with a primary outcome is what was reported in the NEJM paper. Below is the unpublished cumulative incidence information.
Time Frame: Time to event
Population: Randomized participants with at least one day of follow-up, per intent to treat
Measure: Number (95% Confidence Interval); unit: cumulative probability of event
Arm/Group | Patient Self-Testing (PST) | High Quality Anticoagulation Management (HQACM)
Number analyzed (Participants) | 1463 | 1452
cumulative probability of event
  Cumulative Incidence at 500 Days | 0.0785 [0.0645 to 0.0925] | 0.0987 [0.0830 to 0.1144]
  Cumulative Incidence at 1000 Days | 0.1542 [0.1349 to 0.1734] | 0.1820 [0.1610 to 0.2031]
  Cumulative Incidence at 1500 Days | 0.2268 [0.2002 to 0.2535] | 0.2524 [0.2229 to 0.2818]
Statistical Analysis 1: Comparison: Patient Self-Testing (PST) vs High Quality Anticoagulation Management (HQACM); The null hypothesis was the hazard ratio was equal to 1; Test type: Non-Inferiority or Equivalence — A target of 363 patients with primary events required to discern a 32% relative drop in annual primary event rates with 90% power (from 5.5% for HQACM to 3.75% for PST) was based on a sample size of 3200 patients with 1 year of enrollment and a minimum of 2 years follow-up. Due to slower than planned enrollment, we randomized 2922 patients over 2.75 years, with a mean follow-up of 3 years; p = 0.14, Log Rank; Hazard Ratio (HR) = 0.88

2. Secondary Outcome: Time in Therapeutic Range Over Full Length of Follow-up (0 to 100 Percent)
Description: Time in target range (TTR) based on Prothrombin Time standardized to the International Normalized Ratio
Time Frame: Full length of follow-up; average of 3 years
Population: Randomized participants with at least one day of follow-up, per intent to treat
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Patient Self-Testing (PST) | High Quality Anticoagulation Management (HQACM)
Number analyzed (Participants) | 1463 | 1452
percentage | 66.2 (14.2) | 62.4 (17.1)

3. Secondary Outcome: DASS at 2 Years of Follow-up
Description: Satisfaction with care was quantified using the Duke Anticoagulation Satisfaction Scale (DASS). Scores range from 25 to 225, with lower scores indicating higher satisfaction.
Time Frame: At two years of follow-up
Population: Randomized participants with at least one day of follow-up, per intent to treat
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Patient Self-Testing (PST) | High Quality Anticoagulation Management (HQACM)
Number analyzed (Participants) | 1120 | 929
score | 46.8 (16.3) | 49.2 (18.0)

4. Secondary Outcome: Cumulative Gain in Health Utilities at 2 Year
Description: Scores range from -0.36 to 1.00 per year, with a negative score indicating a state worse than being dead and a score of 1.00 indicating perfect health. Since the time frame is 2 years, the range is -0.72 to 2.00.
Time Frame: After 2 years of follow-up for each subject
Population: Randomized participants with at least one day of follow-up, per intent to treat
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Patient Self-Testing (PST) | High Quality Anticoagulation Management (HQACM)
Number analyzed (Participants) | 1183 | 997
score | 1.204 (0.619) | 1.049 (0.575)

5. Secondary Outcome: Health Care Costs at 2 Year
Time Frame: After 2 years of follow-up for each subject
Population: Randomized participants with at least one day of follow-up, per intent to treat
Measure: Mean (Standard Deviation); unit: U.S. Dollars
Arm/Group | Patient Self-Testing (PST) | High Quality Anticoagulation Management (HQACM)
Number analyzed (Participants) | 1463 | 1452
U.S. Dollars | 25,754 (35,673) | 24,505 (31,827)

ADVERSE EVENTS:
Time Frame: Full length of follow-up
Description: Serious Adverse Events (SAEs) and non-serious AEs were coded using the Medical Dictionary for Regulatory Activities (MedDRA) version 6.1. The verbatim description was used to classify events by Body System affected (System Organ Class or SOC) and to group using a common medical term (Preferred Term or PT).
Arm/Group | Patient Self-Testing (PST) | High Quality Anticoagulation Management (HQACM)
Serious Adverse Events (participants affected / at risk) | 247/1465 | 250/1457
Other Adverse Events (participants affected / at risk) | 399/1465 | 332/1457
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patient Self-Testing (PST) (N=1465) | High Quality Anticoagulation Management (HQACM) (N=1457)
Abdominal aortic aneurysm (Vascular disorders) | 0 (0) | 1 (1)
Abdominal hematoma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Acute leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Acute myeloid leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Anoxic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Aortic aneurysm rupture (Vascular disorders) | 1 (1) | 0 (0)
Aortic dissection (Vascular disorders) | 0 (0) | 1 (1)
ARDS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Arterial embolism limb (Vascular disorders) | 1 (1) | 0 (0)
Arterial hemorrhage (Vascular disorders) | 0 (0) | 1 (1)
Arteriosclerotic cardiovascular disease (Vascular disorders) | 3 (3) | 0 (0)
Arteriovenous fistula site bleeding (Injury, poisoning and procedural complications) | 0 (0) | 1 (4)
Arteriovenous malformations (Congenital, familial and genetic disorders) | 2 (2) | 2 (3)
Aspiration pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Asystole (Cardiac disorders) | 0 (0) | 1 (1)
Atherosclerotic cardiovascular disease (Vascular disorders) | 2 (2) | 3 (3)
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bleeding (Vascular disorders) | 1 (1) | 0 (0)
Bleeding esophageal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Bleeding gastric ulcer (Gastrointestinal disorders) | 2 (2) | 1 (1)
Bleeding intracranial (Nervous system disorders) | 1 (1) | 0 (0)
Blood clot in urine (Renal and urinary disorders) | 1 (2) | 0 (0)
Bowel infarction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Brain herniation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Brain stem hemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Brain tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Carcinoma duodenum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Carcinoma vocal cord (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 4 (4) | 3 (3)
Cardiac arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac death (General disorders) | 1 (1) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac ischemia (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac procedure complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cardiac valve replacement complication (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 2 (2) | 0 (0)
Cardiopulmonary arrest (Cardiac disorders) | 2 (2) | 1 (1)
Cardiovascular collapse (Vascular disorders) | 1 (1) | 0 (0)
Cellulitis of hand (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis of leg (Infections and infestations) | 1 (1) | 0 (0)
Cerebellar hemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral hematoma (Nervous system disorders) | 2 (2) | 1 (1)
Cerebral hemorrhage (Nervous system disorders) | 1 (1) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 7 (9) | 10 (10)
"Chronic ischemic heart disease, unspecified" (Cardiac disorders) | 0 (0) | 1 (1)
Chronic lymphocytic leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Chronic renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Chronic subdural hematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Collapse of lung (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Congestive heart failure (Cardiac disorders) | 11 (11) | 14 (14)
COPD (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 5 (5)
COPD exacerbation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cor pulmonale (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery bypass (Surgical and medical procedures) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 2 (2)
Coronary artery occlusion (Cardiac disorders) | 1 (1) | 0 (0)
Death (General disorders) | 22 (22) | 19 (19)
Deep vein thrombosis (Vascular disorders) | 1 (2) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dissecting aortic aneurysm (Vascular disorders) | 0 (0) | 1 (1)
Diverticulitis intestinal hemorrhagic (Gastrointestinal disorders) | 4 (4) | 1 (1)
Diverticulum intestinal hemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Drug interaction (General disorders) | 0 (0) | 1 (1)
Duodenal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Embolic stroke (Nervous system disorders) | 2 (3) | 0 (0)
Embolus (Vascular disorders) | 1 (1) | 0 (0)
End stage heart disease (Cardiac disorders) | 0 (0) | 1 (1)
Endocarditis (Infections and infestations) | 1 (1) | 0 (0)
Endocarditis staphylococcal (Infections and infestations) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (3)
Esophageal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Esophageal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Explosion injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Eye hemorrhage (Eye disorders) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Femoral artery occlusion (Vascular disorders) | 0 (0) | 1 (1)
Gastric bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastroesophageal junction ulcer (Gastrointestinal disorders) | 0 (0) | 1 (2)
Gastrointestinal ulcer bleeding (Gastrointestinal disorders) | 0 (0) | 4 (4)
GI bleed (Gastrointestinal disorders) | 24 (30) | 33 (50)
Gum bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Heart failure (Cardiac disorders) | 0 (0) | 5 (5)
Hemarthrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Hematoma (Vascular disorders) | 6 (6) | 4 (4)
Hematoma muscle (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Hematuria (Renal and urinary disorders) | 1 (1) | 5 (5)
Hematuria traumatic (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Hemopneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Hemorrhage intraperitoneal (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hemorrhagic shock (Vascular disorders) | 1 (1) | 0 (0)
Hemorrhagic stroke (Nervous system disorders) | 1 (1) | 1 (1)
Hemorrhagic transformation stroke (Nervous system disorders) | 0 (0) | 1 (1)
Hemorrhagic tumor necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hemorrhoidal bleeding (Gastrointestinal disorders) | 2 (2) | 1 (1)
Hemothorax (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hepatorenal syndrome (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hodgkin*s lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hyphema (Eye disorders) | 0 (0) | 1 (1)
Hypoxic brain damage (Nervous system disorders) | 0 (0) | 1 (1)
Incision site bleeding (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Incision site haematoma (Injury, poisoning and procedural complications) | 1 (1) | 2 (3)
Infectious diarrhea (Infections and infestations) | 1 (1) | 0 (0)
Inflammatory bowel disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intracerebral hemorrhage (Nervous system disorders) | 1 (1) | 1 (1)
Intracranial hematoma (Nervous system disorders) | 1 (1) | 1 (1)
Intracranial hemorrhage (Nervous system disorders) | 3 (3) | 1 (1)
Intraoperative bleeding (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ischemic cardiomyopathy (Cardiac disorders) | 1 (1) | 2 (2)
Joint bleeding (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lacunar infarction (Nervous system disorders) | 1 (1) | 0 (0)
Leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Leukemia myelogenous (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
"Liver, cancer of" (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
Lung mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Mallory Weiss tear (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mediastinal hematoma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Mediastinitis (Infections and infestations) | 1 (1) | 0 (0)
Melena (Gastrointestinal disorders) | 1 (1) | 0 (0)
Metastatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastatic disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
"Metastatic neoplasm NOS, primary site unknown" (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Middle cerebral artery stroke (Nervous system disorders) | 1 (1) | 0 (0)
Middle cerebral artery thrombosis (Nervous system disorders) | 1 (1) | 0 (0)
Motor cycling accident (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Motor vehicle accident (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Multi organ failure (General disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 7 (7) | 6 (6)
Neuroendocrine carcinoma of the skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neutropenic sepsis (Infections and infestations) | 1 (1) | 0 (0)
Non-Q wave MI (Cardiac disorders) | 4 (5) | 0 (0)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Nosocomial pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Occult blood positive (Investigations) | 1 (1) | 0 (0)
Pancreatic adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pancreatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Pancreatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pelvic hematoma (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Perforation post colonoscopy (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 5 (5) | 6 (6)
Pneumonia MRSA (Infections and infestations) | 0 (0) | 1 (1)
Polypectomy (Surgical and medical procedures) | 0 (0) | 2 (2)
Portal vein thrombosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Post biopsy bleeding (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Post procedural bleeding (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Postoperative bleeding (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Postoperative complication (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Q wave MI (Cardiac disorders) | 2 (2) | 0 (0)
Radiation esophagitis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Radiation pneumonitis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rectal bleeding (Gastrointestinal disorders) | 3 (3) | 5 (5)
Renal artery aneurysm (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 2 (2) | 0 (0)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (5)
Retinal artery occlusion (Eye disorders) | 1 (1) | 0 (0)
Retinal hemorrhage (Eye disorders) | 1 (1) | 1 (1)
Retroperitoneal bleed (Gastrointestinal disorders) | 0 (0) | 2 (2)
Ruptured appendix (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ruptured cerebral aneurysm (Nervous system disorders) | 1 (1) | 0 (0)
Ruptured diverticulum (Gastrointestinal disorders) | 0 (0) | 1 (1)
Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Scrotal abscess (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 6 (6) | 5 (5)
Septic shock (Infections and infestations) | 1 (1) | 2 (2)
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Stoma site bleeding (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Strangulated hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Subarachnoid hemorrhage (Nervous system disorders) | 1 (1) | 2 (3)
Subdural hematoma (Injury, poisoning and procedural complications) | 2 (2) | 7 (7)
Sudden cardiac death (General disorders) | 1 (1) | 2 (2)
Sudden death (General disorders) | 0 (0) | 1 (1)
Suicide (Psychiatric disorders) | 1 (1) | 1 (1)
Thromboembolism (Vascular disorders) | 0 (0) | 1 (1)
Tongue hematoma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 9 (9) | 9 (10)
Transient ischemic attacks (Nervous system disorders) | 0 (0) | 1 (1)
Traumatic hematoma (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Traumatic hemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
UGI bleed (Gastrointestinal disorders) | 4 (4) | 4 (4)
Unknown primary cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Unspecified disease of respiratory system (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Vascular pseudoaneurysm (Vascular disorders) | 1 (1) | 1 (1)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 2 (2)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 2 (2)
Ventricular tachycardia (Cardiac disorders) | 2 (2) | 0 (0)
Vitreous hemorrhage (Eye disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patient Self-Testing (PST) (N=1465) | High Quality Anticoagulation Management (HQACM) (N=1457)
Abrasions (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Anemia postoperative (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Arteriovenous graft site hemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (4)
Arteriovenous malformation (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Bleeding (Vascular disorders) | 32 (45) | 27 (31)
Bleeding from ears (Ear and labyrinth disorders) | 4 (4) | 7 (7)
Bleeding from tongue (Gastrointestinal disorders) | 1 (1) | 2 (2)
Bleeding gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Bleeding genital (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Bleeding lips (Gastrointestinal disorders) | 0 (0) | 4 (4)
Bleeding mouth (Gastrointestinal disorders) | 5 (5) | 3 (3)
Bleeding urogenital (Renal and urinary disorders) | 1 (1) | 0 (0)
Bleeding varicose vein (Vascular disorders) | 1 (1) | 0 (0)
Blood in stool (Gastrointestinal disorders) | 5 (5) | 5 (5)
Bruising (Injury, poisoning and procedural complications) | 7 (8) | 4 (5)
Catheter site bleeding (General disorders) | 1 (1) | 2 (2)
Catheter site hematoma (General disorders) | 0 (0) | 1 (1)
Cellulitis of finger (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis of leg (Infections and infestations) | 0 (0) | 1 (1)
Central line complication (General disorders) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Circumcision (Surgical and medical procedures) | 0 (0) | 2 (2)
Conjunctival bleeding (Eye disorders) | 4 (4) | 3 (3)
Corneal bleeding (Eye disorders) | 1 (1) | 0 (0)
Cystoscopy (Investigations) | 1 (1) | 0 (0)
Deep venous thrombosis arm (Vascular disorders) | 2 (2) | 2 (2)
Deep venous thrombosis femoral (Vascular disorders) | 1 (1) | 1 (1)
Diverticulosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dog bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
DVT (Vascular disorders) | 2 (2) | 8 (8)
Ecchymosis (Skin and subcutaneous tissue disorders) | 12 (21) | 0 (0)
Effusion pleural bloody (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Embolus arm (Vascular disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 79 (130) | 63 (88)
Eye hemorrhage (Eye disorders) | 1 (1) | 1 (1)
Fecal occult blood (Investigations) | 1 (1) | 0 (0)
Femoral artery injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Foot injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Foot ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Gallbladder hemorrhage (Hepatobiliary disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal arteriovenous malformation (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
GI bleed (Gastrointestinal disorders) | 27 (28) | 18 (19)
Gingival bleeding (Gastrointestinal disorders) | 3 (3) | 7 (7)
Haemorrhagic transformation stroke (Nervous system disorders) | 0 (0) | 1 (1)
Hemarthrosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Hematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hematochezia (Gastrointestinal disorders) | 0 (0) | 3 (3)
Hematoma (Vascular disorders) | 25 (25) | 14 (14)
Hematoma muscle (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Hematospermia (Reproductive system and breast disorders) | 6 (7) | 1 (1)
Hematuria (Renal and urinary disorders) | 67 (89) | 54 (72)
Hemoperitoneum (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 11 (13) | 17 (19)
Hemorrhage from throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Hemorrhagic stroke (Nervous system disorders) | 1 (1) | 2 (2)
Hemorrhagic transformation stroke (Nervous system disorders) | 1 (1) | 1 (1)
Hemorrhoidal bleeding (Gastrointestinal disorders) | 10 (13) | 9 (10)
Hemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Ileostomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Incision site bleeding (Injury, poisoning and procedural complications) | 8 (8) | 3 (3)
Incision site hematoma (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Injection site bleeding (General disorders) | 0 (0) | 2 (2)
Intracardiac thrombus (Cardiac disorders) | 0 (0) | 1 (1)
Intracranial hemorrhage (Nervous system disorders) | 1 (1) | 1 (1)
Intraocular hemorrhage (Eye disorders) | 7 (7) | 2 (2)
Intraoperative bleeding (Injury, poisoning and procedural complications) | 8 (9) | 12 (12)
Joint bleeding (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Joint hematoma (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 19 (20) | 12 (12)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mallory Weiss tear (Gastrointestinal disorders) | 0 (0) | 1 (1)
Melena (Gastrointestinal disorders) | 2 (2) | 2 (2)
Muscle hemorrhage (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Myelodysplasia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 4 (4) | 1 (1)
Non-Q wave MI (Cardiac disorders) | 19 (19) | 18 (18)
Ocular retrobulbar hemorrhage (Eye disorders) | 1 (1) | 0 (0)
Perforation post colonoscopy (Gastrointestinal disorders) | 2 (2) | 0 (0)
Pleural hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Post biopsy bleeding (Injury, poisoning and procedural complications) | 4 (4) | 3 (3)
Post procedural bleeding (Injury, poisoning and procedural complications) | 13 (13) | 7 (9)
Postoperative bleeding (Injury, poisoning and procedural complications) | 9 (9) | 15 (15)
Postoperative hematoma (Injury, poisoning and procedural complications) | 5 (5) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (5)
Q wave MI (Cardiac disorders) | 2 (2) | 3 (3)
Rectal bleeding (Gastrointestinal disorders) | 32 (39) | 35 (40)
Renal artery embolism (Renal and urinary disorders) | 0 (0) | 1 (1)
Respiratory tract hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Retinal vein occlusion (Eye disorders) | 0 (0) | 1 (1)
Retroperitoneal bleed (Gastrointestinal disorders) | 8 (10) | 4 (4)
Scleral hemorrhage (Eye disorders) | 2 (2) | 2 (2)
Scrotal hematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Scrotal hemorrhage (Reproductive system and breast disorders) | 2 (2) | 1 (1)
Stroke (Nervous system disorders) | 24 (29) | 34 (41)
Subconjunctival hemorrhage (Eye disorders) | 10 (11) | 2 (2)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Testicular hemorrhage (Reproductive system and breast disorders) | 1 (2) | 0 (0)
Traumatic hematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
UGI bleed (Gastrointestinal disorders) | 4 (4) | 5 (6)
Urethral hemorrhage (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary tract bleeding (Renal and urinary disorders) | 8 (11) | 9 (9)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Venous injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vitreous hemorrhage (Eye disorders) | 0 (0) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes